CLINICAL TRIAL: NCT00505115
Title: The Human Blastocyst Secretome and Implantome
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Other Study IDs: VLC-CS-0707-707-30
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2007-07

CONDITIONS: Blastocyst

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to identify the protein secretion and consumption profile of the human blastocyst (secretome) and the implanted blastocyst (implantome) using the protein array technology.

ELIGIBILITY:
Inclusion Criteria:

* Conditioned medium of blastocytes

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simon, MD PhD, Principal Investigator — Fundación para la Investigación del Instituto Valenciano de Infertilidad (FIVI)
Locations (1):
- Fundación para la Investigación del Instituto Valenciano de Infertilidad (FIVI), Valencia, Valencia, Spain